CLINICAL TRIAL: NCT02119858
Title: A Prospective Investigation of Near Infrared Fluorescence Imaging of Pelvic Lymph Nodes Using Indocyanine Green on the da Vinci Surgical System During Radical Prostatectomy and Pelvic Lymphadenectomy for Localized Prostate Cancer
Brief Title: Diffuse Optical Imaging With Indocyanine Green Solution in Imaging Pelvic Lymph Nodes in Patients With Stage II Prostate Cancer Undergoing Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14015; NCI-2014-00711 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14015 (Other: City of Hope Medical Center)
Record Dates: First submitted 2014-04-09; First posted 2014-04-22 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Stage IIA Prostate Cancer; Stage IIB Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (ICG, diffuse optical imaging, surgery) (Experimental): Patients receive indocyanine green transperineally and undergo diffuse optical imaging during robot-assisted laparoscopic radical prostatectomy with bilateral lymph node dissection using the da Vinci Robotic Surgical System.
  Interventions: Drug: indocyanine green solution; Other: diffuse optical imaging; Procedure: robot-assisted laparoscopic surgery; Procedure: therapeutic lymphadenectomy

INTERVENTIONS:
Drug: indocyanine green solution — Given transperineally
  Other Names: IC-GREEN; ICG solution
Other: diffuse optical imaging — Undergo near infrared fluorescence imaging
  Other Names: diffuse optical spectroscopy; diffuse optical tomography; DOI; near infrared optical tomography
Procedure: robot-assisted laparoscopic surgery — Undergo robot-assisted laparoscopic radical prostatectomy
Procedure: therapeutic lymphadenectomy — Undergo lymphadenectomy

SUMMARY:
This clinical trial studies diffuse optical imaging with indocyanine green solution in imaging pelvic lymph nodes in patients with stage II prostate cancer undergoing surgery. Indocyanine green solution is a special dye that can help doctors see the lymph nodes and blood vessels during surgery when visualized under diffuse optical imaging. Indocyanine green solution may improve the ability to detect lymph nodes and may lead to improved accuracy of lymph node removal.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the ability of indocyanine green (indocyanine green solution) (ICG) to highlight pelvic lymphatic tissue with fluorescence during robot assisted radical prostatectomy using near infrared fluorescence (diffuse optical imaging).

SECONDARY OBJECTIVES:

I. To evaluate the ability of this technique to improve lymph node yield, providing a potential therapeutic benefit to these patients by removing additional lymph nodes that may otherwise have been missed.

OUTLINE:

Patients receive indocyanine green transperineally and undergo diffuse optical imaging during robot-assisted laparoscopic radical prostatectomy with bilateral lymph node dissection using the da Vinci Robotic Surgical System.

After completion of study treatment, patients are followed up for 1-2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Stage 2, intermediate to high risk (per D'Amico criteria) localized prostate cancer with a prostate gland size =< 100 grams

  * Intermediate risk: prostate specific antigen (PSA) between 10-20, Gleason grade 7, or clinical stage T2b
  * High risk: PSA > 20 , Gleason grade >= 8, or clinical stage >= T2c
* Life expectancy of at least 10 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* The subject must be able to comply with the study procedures
* All subjects must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Subject has significant liver disease, cirrhosis or liver insufficiency with abnormal liver function tests, as total bilirubin > 1.5 x normal
* Subject has significant liver disease, cirrhosis or liver insufficiency with abnormal liver function tests, as serum glutamic oxaloacetic transaminase (SGOT) > 2 x normal
* Prior prostate surgery (i.e. transurethral resection of the prostate), or any prior abdominal or pelvic surgery, most specifically for surgeries that may have included any form of lymphadenectomy or anatomic changes
* History of androgen deprivation therapy, any prior chemotherapy, or any prior radiation therapy to the pelvis
* Subject has a previous history of adverse reaction or allergy to ICG, iodine, shellfish or iodine dyes
* Subject in whom the use of x-ray dye or ICG is contraindicated including development of adverse events when previously or presently administered
* Subject has any medical condition, which in the judgment of the investigator and/or designee makes the subject a poor candidate for the investigational procedure
* The presence of medical conditions contraindicating general anesthesia or standard surgical approaches

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07-25; Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

PRIMARY OUTCOMES:
Intraoperative detection of fluorescence in pelvic lymphatic tissue by near-infrared imaging technology on the da Vinci Surgical System following direct injection of ICG into the prostate | At the time of surgery
  The ability to image lymph nodes prior to dissection will be estimated using means and standard errors for all observations as well as stratified by dose level and other relevant patient characteristics.

SECONDARY OUTCOMES:
Quality of fluorescence as detected by near-infrared technology on the da Vinci Surgical System of lymphatic tissue at varying safe doses of ICG | At the time of surgery
  Analyzed using means and standard errors for continuous data and generating frequencies and percentages for categorical data. The Kruskal Wallis test and chi-square test (or Fisher's exact test as appropriate) will be used to detect any apparent differences in continuous and categorical data, respectively.
Lymph node yield | At the time of surgery
  Analyzed using means and standard errors for continuous data and generating frequencies and percentages for categorical data. The Kruskal Wallis test and chi-square test (or Fisher's exact test as appropriate) will be used to detect any apparent differences in continuous and categorical data, respectively.
Number of positive lymph nodes (nodes that contain cancer on final pathology) | At the time of surgery
  Analyzed using means and standard errors for continuous data and generating frequencies and percentages for categorical data. The Kruskal Wallis test and chi-square test (or Fisher's exact test as appropriate) will be used to detect any apparent differences in continuous and categorical data, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Bertram Yuh, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States